CLINICAL TRIAL: NCT00288483
Title: Placebo-Controlled, Randomised, Double-Blind, Multi-Centre Clinical Trial on Dose-Dependent Cholesterol-Lowering Effects of Policosanol in Patients With Hypercholesterolaemia With 10 to 80 Mg Policosanol for 12 Weeks
Brief Title: Cholesterol-Lowering Effects of Policosanol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Drug Commission of the German Medical Association (Other)
Collaborators: Madaus AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC53W0.01
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-11

CONDITIONS: Hypercholesterolemia; Combined Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — policosanol

INTERVENTIONS:
Drug: Policosanol

SUMMARY:
Despite undeniable progress in the reduction of morbidity and mortality of coronary heart disease (CHD) prevention is a mainstay for medical intervention. The importance of elevated serum cholesterol for the formation and progress of CHD can be regarded as proved after the results of the major intervention studies became available. These studies have provided key evidence for a positive correlation of lipid lowering and decreased mortality. Other studies in patients with established CHD have shown that stabilization and regression of atherosclerotic lesions is possible with lowering of cholesterol using a variety of agents. Different studies have also investigated the long-term effects of lipid lowering strategies on atherosclerosis by means of coronary angiography and have demonstrated that lipid reduction reduces progression of atherosclerosis and can promote atherosclerosis regression. Thus, it has been demonstrated that cholesterol lowering therapy reduces the risk of CHD and diminishes cardiovascular morbidity and mortality.

Policosanol is a drug that presumably possesses both hypocholesterolemic and antiplatelet effects. Furthermore there are hints to even more positive effects that influence the development of atherosclerosis, i.e. inhibition of LDL peroxidation and smooth muscle cell proliferation.

Previous studies showed efficacy in dose ranges of mostly 5 to 20 mg Policosanol per day. As nearly all previous studies have been performed in Latin America it cannot be excluded that either ethnic or nutritional factors contribute to the dose found to be optimal in this region. This circumstance as well as the requirement to meet the ICH Guideline "Ethnic Factors in the Acceptability of Foreign Clinical Data" make further studies, i.e. a dose-finding clinical trial, an efficacy clinical trial in European patients and a long-term tolerability clinical trial in Caucasian patients necessary.

It is known from more than 60 clinical studies performed so far that Policosanol has an excellent safety profile. A placebo-controlled design was considered appropriate as patients with two or more risk factors for the development of cardiovascular events and a LDL of greater than 190 mg/dl were excluded; the chance of getting an active lipid-lowering agent during the treatment phase was 80 %.

DETAILED DESCRIPTION:
Visit 1: Informed consent, Inclusion and exclusion criteria, medical history, concomitant diseases and medication, physical examination, vital signs, lipid profile, safety lab, urine analysis, 12-lead EKG. Diet counseling.

Run-in phase six weeks. Visit 2 and 3 (5 and 6 weeks after visit 1): Baseline lipids. Visit 4: Baseline lipid sample, start treatment. Randomization to one of five groups, placebo, 10 mg, 20 mg, 40 mg, or 80 mg policosanol.

Visit 5 and 6 (6 and 12 weeks after visit 4): Lipid sample. Safety lab.

ELIGIBILITY:
Inclusion Criteria:

* Isolated hypercholesterolaemia or combined hyperlipidaemia with mean LDL values at Visits 2 and 3 of > 150 mg/dl for patients with no or one risk factor (other than known coronary artery disease) or 150-189 mg/dl for patients with two or more risk factors for the development of cardiovascular events (males > 45 years of age, females > 55 years of age or postmenopausal), known coronary artery disease, uncontrolled hypertension > 140 mm Hg systolic, HDL level < 35 mg/dl (mean of the values of visits 2 and 3), current cigarette smoking of > 10 cigarettes/day, obesity with BMI > 30 kg/m², family history of coronary heart disease),
* male or female patients aged from 18 to 80 years,
* negative pregnancy test for woman of childbearing potential,
* no communication problems with the investigator,
* availability of a signed informed consent to participate in the trial, for medical data to be recorded and made available to a third party.

Exclusion Criteria:

* - known hypersensitivity to any component of the drug,
* myocardial infarction less than one year before clinical trial inclusion,
* PTCA or CABG less than one year before clinical trial inclusion,
* unstable angina pectoris,
* hypothyroidism,
* diabetes mellitus,
* acute inflammatory diseases,
* severe gastrointestinal diseases,
* triglycerides values > 500 mg/dl at Visit 2 or 3,
* use of oral systemic corticosteroids, anticoagulants or other lipid-lowering drugs,
* serious diseases or circumstances not allowing the patient's participation in the trial (e.g. malignoma, alcoholism or drug abuse, severe kidney and liver diseases),
* pregnancy, lactation and women of childbearing potential without employing a safe contraception method,
* participation in a clinical trial within the last 30 days before Visit 1,
* repeated inclusion in the present clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2001-07

PRIMARY OUTCOMES:
Decrease in LDL cholesterol

SECONDARY OUTCOMES:
Changes in other lipoproteins

CONTACTS AND LOCATIONS:
Overall Officials: Heiner K. Berthold, MD, PhD, Principal Investigator — Drug Commission of the German Medical Association

REFERENCES:
- [Result] Berthold HK, Unverdorben S, Degenhardt R, Bulitta M, Gouni-Berthold I. Effect of policosanol on lipid levels among patients with hypercholesterolemia or combined hyperlipidemia: a randomized controlled trial. JAMA. 2006 May 17;295(19):2262-9. doi: 10.1001/jama.295.19.2262. PMID 16705107